CLINICAL TRIAL: NCT01896284
Title: Phase IV Study to Evaluate the Efficacy of Aflibercept in Subjects With Neovascular Age-related Macular Degeneration (wAMD), Without Optimal Response to Repeated Monthly Intravitreal Injections of Anti Vascular Endothelial Growth Factor (Anti VEGF-A) Therapy.
Brief Title: Study to Evaluate Efficacy of Aflibercept in Neovascular Age-related Macular Degeneration Patients Non Responders to Anti-Vascular Endothelial Growth Factor
Acronym: MACBETH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barcelona Macula Foundation (Other)
Collaborators: TFS Trial Form Support (Industry); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMF-AFLI-2013-01; 2013-000848-26 (EudraCT Number)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2018-11-23 (Actual); Status verified 2015-07

CONDITIONS: Wet Macular Degeneration
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.5mg AFLIBERCEPT injection (Experimental): Patients will receive intravitreal injection of aflibercept 0.5mg at baseline, week 4,8,16,24 and 32. Optionally, if intra or subretinal fluid persists at week 12, patients will receive an additional injection.
  Interventions: Drug: 0.5mg aflibercept

INTERVENTIONS:
Drug: 0.5mg aflibercept — 0.5mg aflibercept intravitreal injection will be performed every 4 weeks from baseline to week 8 (3 doses) and every 8 weeks until week 32.
  Other Names: EYLEA

SUMMARY:
Patients with neovascular age-related macular degeneration who do not respond to usual treatment with conventional medications may respond to a new drug of the same class which is designed to block a larger fraction of proangiogenic factors.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men and women ≥ 50 years of age.
* Any choroidal neovascular membranes (CNVM) lesion (occult, minimally classic or classic) secondary to age-related macular degeneration
* Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity of: 20/32 to 20/320 (letter score of 73 to 25) in the study eye.
* Able to return for ALL clinic visits and complete all study-related procedures.
* Absence of other ocular diseases that could affect visual acuity.
* Patients without optimal response to ranibizumab or bevacizumab defined as:

  * Patient with significant persistent or recurrent fluid (intraretinal or subretinal) on OCT or any leakage on fluorescein angiography despite at least 4 injections within last 6 months, being the last OCT with presence of fluid within the 6 weeks after last treatment with ranibizumab or bevacizumab.
  * Patient with significant persistent or recurrent fluid (intraretinal or subretinal) on OCT or any leakage on fluorescein angiography despite three monthly treatment with ranibizumab or bevacizumab.

Exclusion Criteria:

* No scar, fibrosis, or atrophy involving the center of the fovea
* No retina pigment epithelium (RPE) rip/tear involving the central fovea
* Participation in another simultaneous interventional clinical trial
* Prior treatment with anti-VEGF or steroids therapy in the study eye within 28 days of baseline
* Prior treatment with photodynamic therapy (PDT)
* Intraocular surgery (including cataract surgery) in the study eye within 2 months preceding Baseline
* History of vitrectomy surgery, submacular surgery, or other surgical intervention for AMD in the study eye
* Active intraocular inflammation in the study eye
* History of cerebral vascular accident, myocardial infarction, transient ischemic attacks within 3 months of study enrollment.
* Unable to undergo fluorescein angiography or fundus photography because of uncontrolled allergies

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with no fluid on Optical Coherence Tomography (OCT) after loading dose of aflibercept | Week 12
  At week 12 an OCT will be performed to evaluate the changes in intra or subretinal fluid and to determine the percentage of patients with no fluid after 3 doses of aflibercept injected on baseline visit, week 4 and week 8.

SECONDARY OUTCOMES:
Changes in best corrected visual acuity (BCVA)after loading dose | week 12
Changes in OCT central foveal thickness after loading dose | week 12
Anatomic and Visual Acuity outcomes maintained during (every 8 weeks) treatment. | week 40
Determine the time to resolution of any intra/sub retinal fluid on OCT | week 4,8,12,24,32,40
Describe safety of this cohort of patients | baseline, week 4, 8, 12, 24, 32 and 40
  Describe the safety of aflibercept in study patients by determining ocular and non ocular adverse events classified according to type, frequency and severity during 40 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Mones, MD PhD, Principal Investigator — Barcelona Macula Foundation; Carlos Juan Donate, MD, Principal Investigator — Hospital San Carlos, Madrid; Marta Suárez de Figueroa, MD, Principal Investigator — Hosipital Universitario Ramon y Cajal; Jose Luis Olea, MD, Principal Investigator — Hospital Son Espases; Francisco Cabrera, MD, Principal Investigator — Hospital Universitario Insular de Canarias; Laura Sarasols, MD, Principal Investigator — Hospital Universitari General de Catalunya; Javier Araiz, MD, Principal Investigator — Instituto Clínico Quirúrgico de Oftalmología de Bilbao; Jose Maria Ruiz-Moreno, MD, Principal Investigator — Hospital Universitario de Albacete; Ignasi Jürgens, MD PhD, Principal Investigator — Institut Catala de Retina
Locations (1):
- Barcelona Macula Foundation, Barcelona, Spain